CLINICAL TRIAL: NCT06648200
Title: Toripalimab and JS004 Combined With Platinum-based Chemotherapy for Relapsed and Extensive-stage Small Cell Lung Cancer: a Single-center, Randomized Trial
Brief Title: Toripalimab and JS004 Combined With Platinum-based Chemotherapy for Relapsed and Extensive-stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-031
Record Dates: First submitted 2024-10-09; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Small Cell Lung Cancer Extensive Stage; Small Cell Lung Cancer Recurrent
Keywords: small cell lung cancer; Toripalimab; JS004; Extensive-stage; Recurrent
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — toripalimab; Etoposide; Platinum

STUDY DESIGN:
Intervention Model Description: All enrolled patients were randomly assigned to one of two groups. Patients in group 1 received toripalimab combined with etoposide and platinum Chemotherapy; patients in group 2 received toripalimab and JS004 combined with etoposide and platinum Chemotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy With Toripalimab Combined With Platinum-based Doublet Chemotherapy (Active Comparator): In this arm, 50 patients with extensive-stage small cell lung cancer or relapsed within more than 6 months after SCLC radical treatment will receive 4 circles of toripalimab combined with platinum-based doublet chemotherapy. Then patients received maintenance treatment with toripalimab until the disease progressed.
  Interventions: Drug: Toripalimab; Drug: Etoposide; Drug: Platinum
- Therapy With Toripalimab and JS004 Combined With Platinum-based Doublet Chemotherapy (Experimental): In this arm, 50 patients with extensive-stage small cell lung cancer or relapsed within more than 6 months after SCLC radical treatment will receive 4 circles of toripalimab and JS004 combined with platinum-based doublet chemotherapy. Then patients received maintenance treatment with toripalimab and JS004 until the disease progressed.
  Interventions: Drug: JS004; Drug: Toripalimab; Drug: Etoposide; Drug: Platinum

INTERVENTIONS:
Drug: JS004 — Specified dose on specified days.
  Other Names: tifcemalimab
  Arms: Therapy With Toripalimab and JS004 Combined With Platinum-based Doublet Chemotherapy
Drug: Toripalimab — Specified dose on specified days.
Drug: Etoposide — Specified dose on specified days.
Drug: Platinum — Specified dose on specified days.

SUMMARY:
For extensive-stage small cell lung cancer (SCLC), platinum-chemotherapy (cisplatin or carboplatin) combined with etoposide as the first-line treatment is recommended. However, the recurrence rate is extremely high after the initial first-line treatment. For those who relapse or progress within more than six minths after the end of the-first-line treatment, chose the current guideline recommendation trearment plan has the poor prognosis. A new immunotherapeutic strategy is needed to achieve better anti-tumor effects. JS004 is a new antibody targeting B and T lymphocyte attenuator (BTLA), which restrains immune cells; function and leads to immune escape of tumor cells. The combination of PD-1 and BTLA antibodies has shown a good therapeutic effect in solid tumors. This trial aims to investigate the efficacy and safety of the therapeutic regimen of toripalimab and JS004 combined with platinum-based doublet chemotherapy in extensive-stage SCLC or relapsed within more than six months after radical treatment SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form;
2. Aged 18 ≥ years;
3. Histological or cytological diagnosis of SCLC by needle biopsy or EBUS, and extensive stage or recurrent confirmed by imageological examinations or relapsed within more than six months after radical treatment SCLC;
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1;
5. Life expectancy is at least 12 weeks;
6. At least 1 measurable lesion according to RECIST 1.1;
7. Patients with good function of other main organs (liver, kidney, blood system, etc.);
8. Fertile female patients must voluntarily use effective contraceptives from the start of the trial to within 30 days after its completion, and urine or serum pregnancy test results within 7 days prior to enrollment are negative;
9. Unsterilized male patients must voluntarily use effective contraception during the trial period and for 30 days after its conclusion.

Exclusion Criteria:

1. Patients with a malignancy other than SCLC within five years prior to the start of this trial;
2. Participants with any unstable systemic disease (including uncontrolled hypertension, severe arrhythmia, etc.);
3. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
4. Participants who are allergic to the test drug or any auxiliary materials;
5. Participants with active hepatitis B, hepatitis C or HIV;
6. Participants with Interstitial lung disease currently;
7. Pregnant or lactating women;
8. Any malabsorption;
9. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
10. Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 60 months
  It is defined as the time (months) from the first administration of drug in this study to the disease progression or death (including any cause of death in the case of no progression) as recorded in CRF, regardless of whether the patient exits from the treatment or receives other anti-cancer treatment before progression.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 30 months
  ORR is defined according to the RECIST v1.1 criteria.
Treatment-related adverse event (TRAE) | Up to 30 months
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.
Overall survival (OS) | up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Health related quality of life (HRQol)：EORTC-QLQ-C30 | up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 , Version 3). EORTC's QLQ-C30 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options.
Health related quality of life (HRQol)：LC13 | up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (LC13, Version 3).The items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.